CLINICAL TRIAL: NCT07173387
Title: Stereotactic Body Radiotherapy and NALIRIFOX for Locally Advanced Pancreatic Cancer: A Prospective Clinical Trial
Acronym: RAD-NALIRIFOX
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shandong Cancer Hospital and Institute (Other)
Responsible Party: Principal Investigator, Jinbo Yue, Director of Department Radiation Oncology, Shandong Cancer Hospital and Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SDZLEC2025-364-02
Record Dates: First submitted 2025-09-08; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Pancreatic Cancer
Keywords: NALIRIFOX; liposomal irinotecan; SBRT
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Intervention Model Description: Cohort 1: Patients receive 1 cycle of NALIRIFOX followed by early SBRT, with subsequent NALIRIFOX cycles (up to 10-12 cycles) continuing after the completion of SBRT.
  Cohort 2: Patients receive 6-8 cycles of NALIRIFOX followed by late SBRT, with further NALIRIFOX cycles continuing post-SBRT.
Masking Description: This is an open-label study with no masking applied to participants, investigators, or care providers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early SBRT after NALIRIFOX Treatment (Experimental): Participants in this arm will receive 1 cycle of NALIRIFOX followed by early SBRT. NALIRIFOX will be continued for up to 10-12 cycles after the completion of SBRT.
  Interventions: Drug: NALIRIFOX (liposomal irinotecan-based chemotherapy).; Radiation: Stereotactic Body Radiation Therapy (SBRT).
- Late SBRT after NALIRIFOX Treatment (Experimental): Participants in this arm will receive 6-8 cycles of NALIRIFOX followed by late SBRT. NALIRIFOX will be continued for up to 10-12 cycles after the completion of SBRT.
  Interventions: Drug: NALIRIFOX (liposomal irinotecan-based chemotherapy).; Radiation: Stereotactic Body Radiation Therapy (SBRT).

INTERVENTIONS:
Drug: NALIRIFOX (liposomal irinotecan-based chemotherapy). — NALIRIFOX is a chemotherapy regimen that includes liposomal irinotecan, oxaliplatin, 5-fluorouracil (5-FU), and leucovorin, administered intravenously in 10-12 cycles every two weeks.
Radiation: Stereotactic Body Radiation Therapy (SBRT). — Stereotactic Body Radiation Therapy (SBRT) is a form of high-precision radiation therapy that delivers focused radiation beams to the tumor while minimizing damage to surrounding healthy tissue. In this study, SBRT will be applied in two different timing schedules after NALIRIFOX chemotherapy: early after 1 cycle (Cohort 1) or late after 6-8 cycles (Cohort 2). The total radiation dose will be 25-50 Gy, delivered in 5 fractions.

SUMMARY:
This prospective, multicenter clinical study evaluates the efficacy and safety of NALIRIFOX in combination with Stereotactic Body Radiation Therapy (SBRT) for patients with locally advanced unresectable pancreatic cancer. The primary endpoint is progression-free survival (PFS), with secondary endpoints including objective response rate (ORR), disease control rate (DCR), overall survival (OS), and safety assessment. The study involves two cohorts: Cohort 1 (early SBRT after 1 cycle of NALIRIFOX) and Cohort 2 (late SBRT after 6-8 cycles of NALIRIFOX). A total of 42 participants are expected to be enrolled, with a follow-up period of at least 24 months. This trial aims to provide a novel therapeutic option for this patient population.

DETAILED DESCRIPTION:
The study will assess the combination of NALIRIFOX (a chemotherapy regimen including liposomal irinotecan) and SBRT in patients with locally advanced unresectable pancreatic cancer. NALIRIFOX consists of liposomal irinotecan, oxaliplatin, 5-FU, and leucovorin, administered in 10-12 cycles every two weeks. SBRT will be applied after a variable period of chemotherapy, randomzing either early or late in the treatment course. The study's main endpoint is progression-free survival (PFS), which is the time from the start of treatment to disease progression or death. Secondary endpoints include ORR, DCR, and OS, providing a comprehensive evaluation of the treatment's effectiveness. Furthermore, the safety profile of the combination will be evaluated, focusing on adverse events using the NCI-CTCAE version 5.0. A total of 42 patients will be enrolled, with an expected follow-up duration of 24 months. The study is designed to explore whether this combined modality can improve outcomes for patients.

ELIGIBILITY:
Inclusion Criteria:

Adults aged 18-75 years, both male and female. Histologically or cytologically confirmed locally advanced unresectable pancreatic cancer.

No prior chemotherapy or radiatiotherapy for pancreatic cancer. ECOG performance status of 0-1.

Adequate organ function as defined by the following criteria:

Absolute neutrophil count (ANC) ≥ 1,500/μL Platelet count ≥ 100,000/μL Hemoglobin ≥ 9 g/dL Total bilirubin ≤ 1.5 times the upper limit of normal (ULN) Serum creatinine ≤ 1.5 times the ULN AST/ALT ≤ 2.5 times the ULN Ability to provide written informed consent.

Exclusion Criteria:

Prior history of other malignancies (except for curatively treated non-melanoma skin cancer or other cancers with a 5-year disease-free survival).

Active infections or severe medical conditions that would interfere with the study.

Pregnancy or breastfeeding. Known hypersensitivity to any of the study drugs. History of severe allergic reactions to liposomal formulations. Uncontrolled comorbid conditions (e.g., heart failure, chronic kidney disease, or uncontrolled diabetes).

Participation in other clinical trials involving investigational treatments within 30 days of enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2028-10-01 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival | Up to 24 months
  The primary outcome measure is progression-free survival (PFS), which is defined as the time from the start of treatment to the first occurrence of disease progression or death.

SECONDARY OUTCOMES:
Objective Response Rate | up to 24 months.
  Defined as the percentage of patients who achieve a partial or complete response, measured by tumor shrinkage using RECIST 1.1 criteria.
Disease Control Rate | up to 24 months.
  Defined as the percentage of patients who achieve a complete response, partial response, or stable disease.
Overall Survival | up to 24 months.
  Defined as the time from the start of treatment to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Jinbo Yue, Doctor, Principal Investigator — Shandong Cancer Hospital and Institute
Locations (1):
- Shandong Cancer Hospital and Institute, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wainberg ZA, Melisi D, Macarulla T, Pazo Cid R, Chandana SR, De La Fouchardiere C, Dean A, Kiss I, Lee WJ, Goetze TO, Van Cutsem E, Paulson AS, Bekaii-Saab T, Pant S, Hubner RA, Xiao Z, Chen H, Benzaghou F, O'Reilly EM. NALIRIFOX versus nab-paclitaxel and gemcitabine in treatment-naive patients with metastatic pancreatic ductal adenocarcinoma (NAPOLI 3): a randomised, open-label, phase 3 trial. Lancet. 2023 Oct 7;402(10409):1272-1281. doi: 10.1016/S0140-6736(23)01366-1. Epub 2023 Sep 11. PMID 37708904
- [Background] Wang-Gillam A, Li CP, Bodoky G, Dean A, Shan YS, Jameson G, Macarulla T, Lee KH, Cunningham D, Blanc JF, Hubner RA, Chiu CF, Schwartsmann G, Siveke JT, Braiteh F, Moyo V, Belanger B, Dhindsa N, Bayever E, Von Hoff DD, Chen LT; NAPOLI-1 Study Group. Nanoliposomal irinotecan with fluorouracil and folinic acid in metastatic pancreatic cancer after previous gemcitabine-based therapy (NAPOLI-1): a global, randomised, open-label, phase 3 trial. Lancet. 2016 Feb 6;387(10018):545-557. doi: 10.1016/S0140-6736(15)00986-1. Epub 2015 Nov 29. PMID 26615328
- [Background] Shamsi M, Mohammadi A, Manshadi MKD, Sanati-Nezhad A. Mathematical and computational modeling of nano-engineered drug delivery systems. J Control Release. 2019 Aug 10;307:150-165. doi: 10.1016/j.jconrel.2019.06.014. Epub 2019 Jun 20. PMID 31229474
- [Background] Frampton JE. Liposomal Irinotecan: A Review in Metastatic Pancreatic Adenocarcinoma. Drugs. 2020 Jul;80(10):1007-1018. doi: 10.1007/s40265-020-01336-6. PMID 32557396
- [Background] Janssen QP, van Dam JL, Bonsing BA, Bos H, Bosscha KP, Coene PPLO, van Eijck CHJ, de Hingh IHJT, Karsten TM, van der Kolk MB, Patijn GA, Liem MSL, van Santvoort HC, Loosveld OJL, de Vos-Geelen J, Zonderhuis BM, Homs MYV, van Tienhoven G, Besselink MG, Wilmink JW, Groot Koerkamp B; Dutch Pancreatic Cancer Group. Total neoadjuvant FOLFIRINOX versus neoadjuvant gemcitabine-based chemoradiotherapy and adjuvant gemcitabine for resectable and borderline resectable pancreatic cancer (PREOPANC-2 trial): study protocol for a nationwide multicenter randomized controlled trial. BMC Cancer. 2021 Mar 23;21(1):300. doi: 10.1186/s12885-021-08031-z. PMID 33757440
- [Background] Garcia-Aguilar J, Patil S, Gollub MJ, Kim JK, Yuval JB, Thompson HM, Verheij FS, Omer DM, Lee M, Dunne RF, Marcet J, Cataldo P, Polite B, Herzig DO, Liska D, Oommen S, Friel CM, Ternent C, Coveler AL, Hunt S, Gregory A, Varma MG, Bello BL, Carmichael JC, Krauss J, Gleisner A, Paty PB, Weiser MR, Nash GM, Pappou E, Guillem JG, Temple L, Wei IH, Widmar M, Lin S, Segal NH, Cercek A, Yaeger R, Smith JJ, Goodman KA, Wu AJ, Saltz LB. Organ Preservation in Patients With Rectal Adenocarcinoma Treated With Total Neoadjuvant Therapy. J Clin Oncol. 2022 Aug 10;40(23):2546-2556. doi: 10.1200/JCO.22.00032. Epub 2022 Apr 28. PMID 35483010
- [Background] Mellon EA, Hoffe SE, Springett GM, Frakes JM, Strom TJ, Hodul PJ, Malafa MP, Chuong MD, Shridhar R. Long-term outcomes of induction chemotherapy and neoadjuvant stereotactic body radiotherapy for borderline resectable and locally advanced pancreatic adenocarcinoma. Acta Oncol. 2015 Jul;54(7):979-85. doi: 10.3109/0284186X.2015.1004367. Epub 2015 Mar 3. PMID 25734581
- [Background] de Geus SWL, Eskander MF, Kasumova GG, Ng SC, Kent TS, Mancias JD, Callery MP, Mahadevan A, Tseng JF. Stereotactic body radiotherapy for unresected pancreatic cancer: A nationwide review. Cancer. 2017 Nov 1;123(21):4158-4167. doi: 10.1002/cncr.30856. Epub 2017 Jul 14. PMID 28708929
- [Background] Gurka MK, Collins SP, Slack R, Tse G, Charabaty A, Ley L, Berzcel L, Lei S, Suy S, Haddad N, Jha R, Johnson CD, Jackson P, Marshall JL, Pishvaian MJ. Stereotactic body radiation therapy with concurrent full-dose gemcitabine for locally advanced pancreatic cancer: a pilot trial demonstrating safety. Radiat Oncol. 2013 Mar 1;8:44. doi: 10.1186/1748-717X-8-44. PMID 23452509
- [Background] Goyal K, Einstein D, Ibarra RA, Yao M, Kunos C, Ellis R, Brindle J, Singh D, Hardacre J, Zhang Y, Fabians J, Funkhouser G, Machtay M, Sanabria JR. Stereotactic body radiation therapy for nonresectable tumors of the pancreas. J Surg Res. 2012 May 15;174(2):319-25. doi: 10.1016/j.jss.2011.07.044. Epub 2011 Sep 5. PMID 21937061
- [Background] Polistina F, Costantin G, Casamassima F, Francescon P, Guglielmi R, Panizzoni G, Febbraro A, Ambrosino G. Unresectable locally advanced pancreatic cancer: a multimodal treatment using neoadjuvant chemoradiotherapy (gemcitabine plus stereotactic radiosurgery) and subsequent surgical exploration. Ann Surg Oncol. 2010 Aug;17(8):2092-101. doi: 10.1245/s10434-010-1019-y. Epub 2010 Mar 12. PMID 20224860
- [Background] Herman JM, Chang DT, Goodman KA, Dholakia AS, Raman SP, Hacker-Prietz A, Iacobuzio-Donahue CA, Griffith ME, Pawlik TM, Pai JS, O'Reilly E, Fisher GA, Wild AT, Rosati LM, Zheng L, Wolfgang CL, Laheru DA, Columbo LA, Sugar EA, Koong AC. Phase 2 multi-institutional trial evaluating gemcitabine and stereotactic body radiotherapy for patients with locally advanced unresectable pancreatic adenocarcinoma. Cancer. 2015 Apr 1;121(7):1128-37. doi: 10.1002/cncr.29161. Epub 2014 Dec 23. PMID 25538019
- [Background] Petrelli F, Comito T, Ghidini A, Torri V, Scorsetti M, Barni S. Stereotactic Body Radiation Therapy for Locally Advanced Pancreatic Cancer: A Systematic Review and Pooled Analysis of 19 Trials. Int J Radiat Oncol Biol Phys. 2017 Feb 1;97(2):313-322. doi: 10.1016/j.ijrobp.2016.10.030. Epub 2016 Oct 24. PMID 28068239
- [Background] Qian L, Li Q, Baryeh K, Qiu W, Li K, Zhang J, Yu Q, Xu D, Liu W, Brand RE, Zhang X, Chen W, Liu G. Biosensors for early diagnosis of pancreatic cancer: a review. Transl Res. 2019 Nov;213:67-89. doi: 10.1016/j.trsl.2019.08.002. Epub 2019 Aug 15. PMID 31442419
- [Background] Vincent A, Herman J, Schulick R, Hruban RH, Goggins M. Pancreatic cancer. Lancet. 2011 Aug 13;378(9791):607-20. doi: 10.1016/S0140-6736(10)62307-0. Epub 2011 May 26. PMID 21620466
- [Background] Cai J, Chen H, Lu M, Zhang Y, Lu B, You L, Zhang T, Dai M, Zhao Y. Advances in the epidemiology of pancreatic cancer: Trends, risk factors, screening, and prognosis. Cancer Lett. 2021 Nov 1;520:1-11. doi: 10.1016/j.canlet.2021.06.027. Epub 2021 Jun 30. PMID 34216688